CLINICAL TRIAL: NCT01759147
Title: Case Series to Evaluate Clinical Outcome of Coracoclavicular Ligament Repair Using Autogenous Gracilis Tendon in Endobutton System.
Brief Title: Clinical Outcome of Coracoclavicular Ligament Repair Using Autogenous Gracilis Tendon in Endobutton System.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsingborgs Hospital (Other)
Responsible Party: Principal Investigator, Jonas Nordin, Medical Intern, Helsingborgs Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JNStudy01
Record Dates: First submitted 2012-12-23; First posted 2013-01-02 (Estimated); Last update posted 2013-01-02 (Estimated); Status verified 2012-12

CONDITIONS: Acromioclavicular Joint Dislocation.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): Surgical repair of acromioclavicular dislocation.
  Interventions: Procedure: Surgical treatment of acromioclavicular dislocation.

INTERVENTIONS:
Procedure: Surgical treatment of acromioclavicular dislocation. — Coracoclavicular ligament repair using autogenous gracilis tendon implanted using an endobutton system containing fibrewires and a single transclavicular, transcoracoid bone tunnel.

SUMMARY:
There are many surgical methods available for the treatment of patients with acromioclavicular dislocations. No single method has yet proven to be superior to the others.

The purpose of this study is to evaluate the clinical outcome and complications associated with coracoclavicular ligament repair using autogenous gracilis tendon graft implanted in a single transclavicle transcoracoid bone tunnel. The implantation is performed using an endobutton system that augments the repair with fibrewires.

The investigators will prospecitvely follow 30 patients enrolled in the study.

The hypthesis is that this near anatomical repair of the coracoclavicular ligaments will result in good clinical outcome and few complications.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old.
* Shoulder trauma within last 2 weeks.
* Pain from the acromioclavicular joint.

Exclusion Criteria:

* Chronic or concomitant acromioclavicular joint pathology on injured side.
* Previous acromioclavicular joint dislocation on contralateral side.
* Major shoulder pathology on affected side.
* Mental inability to take part in rehabilitation.
* Non Swedish or English speaking patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Complication | 12 months after surgery.
  * Redislocations.
  * Other local complications, eg. infection.
Disabilities of the Arm, Shoulder and Hand Score | 12 months after surgery.

SECONDARY OUTCOMES:
Constant-Murley Score | 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karl Lunsjö, Ass Prof, Study Director — University of Lund
Locations (1):
- Hospital of Helsingborg, Helsingborg, Skåne County, Sweden

REFERENCES:
- [Background] DeBerardino TM, Pensak MJ, Ferreira J, Mazzocca AD. Arthroscopic stabilization of acromioclavicular joint dislocation using the AC graftrope system. J Shoulder Elbow Surg. 2010 Mar;19(2 Suppl):47-52. doi: 10.1016/j.jse.2009.12.014. PMID 20188268
- [Background] Mazzocca AD, Santangelo SA, Johnson ST, Rios CG, Dumonski ML, Arciero RA. A biomechanical evaluation of an anatomical coracoclavicular ligament reconstruction. Am J Sports Med. 2006 Feb;34(2):236-46. doi: 10.1177/0363546505281795. Epub 2005 Nov 10. PMID 16282577
- [Background] Lee SJ, Nicholas SJ, Akizuki KH, McHugh MP, Kremenic IJ, Ben-Avi S. Reconstruction of the coracoclavicular ligaments with tendon grafts: a comparative biomechanical study. Am J Sports Med. 2003 Sep-Oct;31(5):648-55. doi: 10.1177/03635465030310050301. PMID 12975181
- [Background] Costic RS, Labriola JE, Rodosky MW, Debski RE. Biomechanical rationale for development of anatomical reconstructions of coracoclavicular ligaments after complete acromioclavicular joint dislocations. Am J Sports Med. 2004 Dec;32(8):1929-36. doi: 10.1177/0363546504264637. PMID 15572323
- [Background] Wellmann M, Kempka JP, Schanz S, Zantop T, Waizy H, Raschke MJ, Petersen W. Coracoclavicular ligament reconstruction: biomechanical comparison of tendon graft repairs to a synthetic double bundle augmentation. Knee Surg Sports Traumatol Arthrosc. 2009 May;17(5):521-8. doi: 10.1007/s00167-009-0737-9. Epub 2009 Feb 19. PMID 19225755
- [Background] Yoo YS, Tsai AG, Ranawat AS, Bansal M, Fu FH, Rodosky MW, Smolinski P. A biomechanical analysis of the native coracoclavicular ligaments and their influence on a new reconstruction using a coracoid tunnel and free tendon graft. Arthroscopy. 2010 Sep;26(9):1153-61. doi: 10.1016/j.arthro.2009.12.031. Epub 2010 Apr 22. PMID 20810076
- [Background] Yoo JC, Ahn JH, Yoon JR, Yang JH. Clinical results of single-tunnel coracoclavicular ligament reconstruction using autogenous semitendinosus tendon. Am J Sports Med. 2010 May;38(5):950-7. doi: 10.1177/0363546509356976. Epub 2010 Mar 12. PMID 20228243
- [Background] Debski RE, Parsons IM 4th, Woo SL, Fu FH. Effect of capsular injury on acromioclavicular joint mechanics. J Bone Joint Surg Am. 2001 Sep;83(9):1344-51. doi: 10.2106/00004623-200109000-00009. PMID 11568197